CLINICAL TRIAL: NCT02939248
Title: Differences in the Pharmacokinetic and Pharmacodynamic Profile of Ticagrelor and Its Active Metabolite AR-C124900XX Between Patients With Unstable Angina Pectoris Treated With Crushed Ticagrelor and a Combination of Morphine and Naloxone or Morphine Alone - a Randomized Study
Brief Title: Influence of Naloxone on Ticagrelor Pharmacokinetics and Pharmacodynamics in Patients With Unstable Angina Pectoris on Concomitant Treatment With Morphine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Collegium Medicum w Bydgoszczy (Other)
Responsible Party: Principal Investigator, Jacek Kubica, Prof. Jacek Kubica, MD, PhD, Collegium Medicum w Bydgoszczy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUMK202G
Record Dates: First submitted 2016-10-18; First posted 2016-10-19 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Unstable Angina Pectoris
MeSH Terms: conditions — Angina, Unstable | interventions — Ticagrelor; Morphine; Naloxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Crushed ticagrelor followed by morphine (Active Comparator): crushed ticagrelor 180 mg administered orally followed by morphine 5 mg intravenously
  Interventions: Drug: Crushed ticagrelor followed by morphine
- Crushed ticagrelor, morphine,naloxone (Active Comparator): crushed ticagrelor 180 mg administered orally followed by morphine 5 mg intravenously and naloxone 1 mg orally
  Interventions: Drug: Crushed ticagrelor, morphine,naloxone

INTERVENTIONS:
Drug: Crushed ticagrelor followed by morphine — Crushed ticagrelor (180 mg) followed by morphine 5 mg intravenously
  Other Names: Brilique
  Arms: Crushed ticagrelor followed by morphine
Drug: Crushed ticagrelor, morphine,naloxone — Crushed ticagrelor (180 mg) orally followed by morphine 5 mg intravenously and naloxone 1 mg orally
  Other Names: Brilique
  Arms: Crushed ticagrelor, morphine,naloxone

SUMMARY:
The purpose of this study is to evaluate differences in the pharmacokinetics and pharmacodynamics of ticagrelor and its active metabolite between patients who received ticagrelor and morphine followed by naloxone versus patients treated with ticagrelor and morphine alone for unstable angina pectoris.

DETAILED DESCRIPTION:
According to contemporary guidelines, ticagrelor is a recommended antiplatelet agent in acute coronary syndromes, including unstable angina pectoris. Quick platelet inhibition plays pivotal role in the treatment of acute coronary syndromes. As evidenced in the IMPRESSION study, analgesia with morphine delays platelet inhibition in patients with acute myocardial infarction. On the other hand, the results of the MOJITO study prove that administration of crushed ticagrelor tablets leads to quicker platelet blockage.

Taking the above into consideration, we created a pharmacokinetic/pharmacodynamic study aiming to evaluate differences between patients who received crushed ticagrelor orally followed by either 1) a combination of intravenous morphine and orally administered naloxone or 2) intravenous morphine alone.

The primary study outcome is time needed for ticagrelor and its active metabolite to reach their maximum plasma concentration in each study arm. Secondary outcomes include ticagrelor and AR-C124900XX maximum concentration and the area under the plasma concentration curve for both agents.

Platelet reactivity will be assessed with the Multiplate Analyzer in all study participants at nine predefined time points.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Diagnosis of unstable angina
* Male or non-pregnant female, aged 18-80 years
* Provision of informed consent for angiography and PCI
* GRACE score <140 pts

Exclusion Criteria:

* treatment with ticlopidine, clopidogrel, prasugrel or ticagrelor within 14 days before the study enrollment
* current treatment with morphine or any opioid "mi" receptor agonist
* hypersensitivity to ticagrelor
* current treatment with oral anticoagulant or chronic therapy with low-molecular-weight heparin
* active bleeding
* history of intracranial hemorrhage
* recent gastrointestinal bleeding (within 30 days)
* history of coagulation disorders
* platelet count less than <100 x10^3/mcl
* hemoglobin concentration less than 10.0 g/dl
* history of moderate or severe hepatic impairment
* history of major surgery or severe trauma (within 3 months)
* risk of bradycardic events as judged by the investigator
* second or third degree atrioventricular block during screening for eligibility
* history of asthma or severe chronic obstructive pulmonary disease
* kidney disease requiring dialysis
* manifest infection or inflammatory state
* Killip class III or IV during screening for eligibility
* respiratory failure
* history of severe chronic heart failure (NYHA class III or IV)
* concomitant therapy with strong CYP3A inhibitors (ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazadone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir) or strong CYP3A inducers (rifampicin, phenytoin, carbamazepine, dexamethasone, phenobarbital) within 14 days and during study treatment
* body weight below 50 kg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Time to maximum concentration (tmax) for ticagrelor and AR-C124900XX for ticagrelor+morphine vs ticagrelor+morphine+naloxone arms | 6 hours

SECONDARY OUTCOMES:
Maximum ticagrelor and AR-C124900XX concentration at 6h after administration | 6 hours
Area under the plasma concentration-time curve for ticagrelor (AUC 0-6h) | prior to the initial dose and 15 min, 30 min, 45 min, 1h, 2h, 3h, 4h, 6h post dose
Area under the plasma concentration-time curve for AR-C124900XX (AUC 0-6h) | prior to the initial dose and 15 min, 30 min, 45 min, 1h, 2h, 3h, 4h, 6h post dose
Platelet arbitrary aggregation units/min assessed by Multiple Electrode Aggregometry | prior to the initial dose and 30min, 1h, 2h, 3h, 4h, 6h post dose

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Kubica, MD., PhD., Principal Investigator — Cardiology Department, Dr. A. Jurasz University Hospital
Locations (1):
- Cardiology Department, Dr. A. Jurasz University Hospital, Bydgoszcz, Kuyavian-Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes